CLINICAL TRIAL: NCT02269800
Title: An Efficacy Study of Benzalkonium Chloride Solution Clearing the Oral Colonized Bacterium in Hospitalized Patients With COPD
Brief Title: An Efficacy Study of BCS Clearing the Oral Colonized Bacterium in Hospitalized Patients With COPD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lustre Pharmaceutical Lab Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LST-001
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Benzalkonium chloride solution (Experimental): Tid, for 7 days.
  Interventions: Drug: Benzalkonium chloride solution
- Normal saline (Active Comparator): Tid, for 7 days.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Benzalkonium chloride solution — Tid, 7 days
  Other Names: You Ke Shi
  Arms: Benzalkonium chloride solution
Drug: Normal saline — Tid, 7 days
  Other Names: NS
  Arms: Normal saline

SUMMARY:
The purpose of study is to evaluate the efficacy and safety of Benzalkonium Chloride Solution clearing the oral colonized bacterium in hospitalized patients with COPD.

DETAILED DESCRIPTION:
This a randomized, double-blind, parallel, single-center, exploratory trial. 60 patients will be randomized to two treatments: benzalkonium chloride solution treatment or normal saline treatment.The purpose of study is to evaluate the efficacy and safety of benzalkonium chloride solution clearing the oral colonized bacterium in hospitalized patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

1. COPD patients in hospitalized.
2. Aged from18 to 70 years (including 18 and 70).
3. Patients participating in this trial should sign ICFs.
4. Patients with good understanding, could conduct this study with investigators.

Exclusion Criteria:

1. History of mouthwash allergies, allergic rhinitis or dermatitis.
2. Patients with oral ulcers, severe periodontal disease, oral mucosal lesions or oral cancer, patients received special oral clean.
3. Patients with removable denture.
4. Patients with malignant blood diseases.
5. History of using cytotoxic drugs or biological immunosuppressants ( such as TNF-α inhibitors ).
6. Had used clinical study drugs before 28 days enrollment.
7. Had used clinical study drugs before 28 days enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Aerobic pathogenic bacterial colonization rate in oral airway | Day 7

SECONDARY OUTCOMES:
The improvement of oral status | Day 7
The subjective feeling | Day 7
The incidence of hospital acquired respiratory infections | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Shiyue Li, Professor, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University